CLINICAL TRIAL: NCT02766621
Title: Phase 1, Randomized, Double-blind, Third-party Open Placebo-controlled, Dose Escalating Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Single And Multiple Intravenous And Subcutaneous Doses Of Pf-06823859 In Healthy Subjects
Brief Title: Evaluation Of Safety, Tolerability And Pharmacokinetics Of Single And Multiple Doses Of Compound PF-06823859
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C0251001
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: First in human, Phase 1, Healthy volunteers
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo injection SC/IV (Placebo Comparator): Placebo for injection SC/IV
  Interventions: Drug: Placebo injection SC/IV
- PF-06823859 (Active Comparator): Study Drug being used in the study
  Interventions: Biological: PF-06823859

INTERVENTIONS:
Biological: PF-06823859 — Comparison of different dosages of PF-06823859 to placebo
  Other Names: Study drug
  Arms: PF-06823859
Drug: Placebo injection SC/IV — Comparison of Placebo to different doses of PF-06823859
  Other Names: Placebo
  Arms: Placebo injection SC/IV

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of escalating single and multiple intravenous (IV) infusions and subcutaneous (SC) injections of PF 06823859 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non childbearing potential and male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

1. History of active or latent tuberculosis (TB) regardless of treatment; positive Quantiferon - TB test.
2. Subjects with a history of autoimmune disorders.
3. Subjects with a history of or positive results for any of the following serological tests: Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), anti Hepatitis C antibody (HCVAb) or human immunodeficiency virus (HIV).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs | Dosing through approximately Day 189
  Safety

SECONDARY OUTCOMES:
Apparent Clearance (CL) of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Number of Participants With Anti-Drug Antibody (ADA) to PF-06823859 | Pre dose to approximately Day 189
  Immunogenicity
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Maximum Observed Plasma Concentration (Cmax) of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Plasma Decay Half-Life (t1/2) | Pre dose to approximately Day 189
  Pharmacokinetics
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06823859 administered subcutaneously | Pre dose to approximately Day 189
  Pharmacokinetics
Volume of Distribution at Steady State (Vss) of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
AUCtau (dose normalized) | Pre dose to approximately Day 189
  Pharmacokinetics
C av of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Mean residence of time for PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
Maximum Observed Plasma Concentration (Cmax) dose normalized of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics
bioavailability of PF-06823859 subcutaneous doses compared to intravenous doses of PF-06823859 | Pre dose to approximately Day 189
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Neelakantan S, Oemar B, Johnson K, Rath N, Salganik M, Berman G, Pelletier K, Cox L, Page K, Messing D, Tarabar S. Safety, Tolerability, and Pharmacokinetics of PF-06823859, an Anti-Interferon beta Monoclonal Antibody: A Randomized, Phase I, Single- and Multiple-Ascending-Dose Study. Clin Pharmacol Drug Dev. 2021 Mar;10(3):307-316. doi: 10.1002/cpdd.887. Epub 2020 Dec 22. PMID 33352008
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0251001&StudyName=Phase+1%2C+Randomized%2C+Double-blind%2C+Third-party+Open+Placebo-controlled%2C+Dose+Escalating+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+Pharmacokinetics+And+Pharmacodynamics+Of+Single+And+Multiple+Intravenous++And+Subcutaneous+Doses+Of+Pf-06823859+In+Healthy+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C0251001&StudyName=Phase+1%2C+Randomized%2C+Double-blind%2C+Third-party+Open+Placebo-controlled%2C+Dose+Escalating+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+Pharmacokinetics+And+Pharmacodynamics+Of+Single+And+Multiple+Intravenous+And+Subcutaneous+Doses+Of+Pf-06823859+In+Healthy+Subjects